CLINICAL TRIAL: NCT06499805
Title: Barriers and Facilitators to OTC Hearing Aids Success
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Hsiang Wu (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Vanderbilt University Medical Center (Other); University of Manchester (Other)
Responsible Party: Sponsor-Investigator, Yu-Hsiang Wu, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202404595; R01DC015997 (NIH)
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss, Sensorineural; Presbycusis
MeSH Terms: conditions — Hearing Loss, Sensorineural; Presbycusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AUD (audiologist-based) (Active Comparator): In this group, the audiologist-based fitting will be used to provide prescription hearing aids.
  Interventions: Device: Audiologist-based fitting
- OTC (over-the-counter) (Experimental): In this group, over-the-counter fitting will be used to provide over-the-counter hearing aids.
  Interventions: Device: Over-the-counter fitting

INTERVENTIONS:
Device: Audiologist-based fitting — Description hearing aids will be fitted by audiologists using established procedures.
  Arms: AUD (audiologist-based)
Device: Over-the-counter fitting — In this group, over-the-counter hearing aids will be used by subjects. Subjects will take the full initiative and responsibility for learning and using hearing aids.
  Arms: OTC (over-the-counter)

SUMMARY:
Hearing aids can improve hearing, communication, and overall quality of life for people with hearing loss. However, not many people use hearing aids. A common reason is that hearing aids are expensive and hard to get. The traditional way to get hearing aids involves multiple visits to licensed audiologists for identifying hearing loss, customizing the aids, and ongoing maintenance. This traditional method is called the AUD pathway.

Over-the-counter (OTC) hearing aids offer a different approach. They aim to make hearing aids more affordable and accessible, encouraging earlier use. In the OTC pathway, users diagnose their own hearing loss and fit and program the hearing aids themselves. Little is known about long-term effects of OTC hearing aids on users.

This study aims to compare the experiences of people who choose the OTC pathway with those who choose the AUD pathway. It takes place in two locations: Iowa City, IA, and Nashville, TN. Participants, who have mild-to-moderate hearing loss, choose their preferred pathway and are followed for 12 months. In the OTC pathway, participants buy their hearing aids directly from OTC companies or retailers. In the AUD pathway, prescription hearing aids and fitting services are provided by audiology clinics at the University of Iowa and Vanderbilt University Medical Center.

Participants are contacted 1, 6, and 12 months after starting to use their hearing aids. Researchers measure their satisfaction about hearing aids and other outcomes. If participants stop using their hearing aids, researchers assess their engagement with post-amplification hearing care. The results from both pathways are then compared.

DETAILED DESCRIPTION:
Although hearing aids (HAs) can improve hearing ability, communication, social and emotional function, and quality of life for people with hearing loss, the adoption rate of HAs is low. A commonly reported barrier to HA uptake is that HAs are not affordable or accessible under the traditional service delivery model, which requires multiple visits to licensed audiologists for identification of hearing loss, customization of the HAs, and continual maintenance and fine-tuning. This hearing healthcare pathway is referred to as the AUD pathway. As an alternative, over-the-counter (OTC) HAs aim to promote earlier HA adoption and improve HA affordability and accessibility. In this healthcare pathway, referred to as the OTC pathway, users self-diagnose hearing loss and fit and program their OTC HAs. Although prior research has supported the feasibility of HA self-fitting and the OTC service-delivery model, little is known about how the OTC pathway impacts users' long-term well-being.

The goal of this study is to characterize the patient journey of individuals who opt for the OTC pathway in comparison to those who select the AUD pathway. The study is a two-site (Iowa City, IA, and Nashville, TN) longitudinal study in which participants choose their preferred healthcare pathways (OTC vs. AUD), and their HA outcomes are tracked for 12 months. Adults with bilateral mild-to-moderate hearing loss are recruited from the community. Upon entering the study, participants choose their preferred pathway and then proceed with the purchase of HAs. In the OTC pathway, participants purchase their chosen OTC HAs directly from OTC companies or retailers. In the AUD pathway, prescription HAs and fitting services are offered by the audiology clinics at the University of Iowa and Vanderbilt University Medical Center. Participants are contacted 1, 6, and 12 months after they begin using their HAs. During each contact, HA outcomes (e.g., HA satisfaction) are measured if participants continue using HAs. If participants have abandoned or under-utilized their HAs, their engagement with post-amplification hearing healthcare behaviors (e.g., seeking HAs again) is assessed. The data from the OTC and AUD pathways are then compared.

ELIGIBILITY:
Inclusion Criteria:

* adult-onset, perceived bilateral mild-to-moderate hearing loss
* no previous hearing aid experience

Exclusion Criteria:

* Non-native speaker of English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Hearing aid satisfaction as measured by the Satisfaction with Amplification in Daily Life (SADL) | 1-, 6-, and 12-month post-intervention
  The SADL is a questionnaire designed to measures subject's perceived hearing aid satisfaction. The score ranges from 1 (low satisfaction) to 7 (high satisfaction).

SECONDARY OUTCOMES:
Overall hearing aid outcome as measured by the International Outcome Inventory for Hearing Aids (IOI-HA) | 1-, 6-, and 12-month post-intervention
  The IOI-HA is a questionnaire designed to measures hearing aid outcome across multiple domains, including hearing aid use time and satisfaction. The score ranges from 1 (poor outcome) to 5 (great outcome).
Aided hearing-specific quality of life as measured by the the Revised Hearing Handicap Inventory (RHHI). | 1-, 6-, and 12-month post-intervention
  The RHHI is designed to measure subject's hearing-specific quality of life (i.e., perceived hearing handicap). The score ranges from 0 (no handicap) to 24 (more handicap).
Hearing aid related issues as measured by the Hearing Aid Issues Survey | 1-, 6-, and 12-month post-intervention
  This questionnaire asks participants to report the frequency of occurrence of 15 common device-related issues (e.g., "whistles", "device hurts ear", and ?too loud?) using a 5-point Likert scale. The score ranges from 15 (no issues) to 75 (more issue).
Hearing aid success as measured by the HA Use Questionnaire | 1-, 6-, and 12-month post-intervention
  This instrument has three hearing aid use patterns to choose from: full-time use (whenever hearing aids are needed, score=3), part-time use (occasional use, score=2), and non-use (score=1).
Engagement with post-amplification hearing healthcare behaviors measured by the Hearing Healthcare Behavior Questionnaire | 1-, 6-, and 12-month post-intervention
  This questionnaire measures the participants' engagement with hearing healthcare behaviors after they have abandoned or under-utilized the study HAs (e.g., seeking HAs again). The score ranges from 0 (no engagement) to 1 (full engagement).

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Wu, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from a total of 360 participants with hearing loss recruited State of Iowa, State of Tennessee and surrounding areas. The final dataset will include self-reported hearing aid outcome data. All datasets and metadata that can be shared will be deposited in the Inter-University Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available no later than the publication of the main findings.
Access Criteria: The data will be deposited in the Inter-University Consortium for Political and Social Research (ICPSR), and will be available to the public.

REFERENCES:
- [Background] Brody L, Wu YH, Stangl E. A Comparison of Personal Sound Amplification Products and Hearing Aids in Ecologically Relevant Test Environments. Am J Audiol. 2018 Dec 6;27(4):581-593. doi: 10.1044/2018_AJA-18-0027. PMID 30458521
- [Background] Chien W, Lin FR. Prevalence of hearing aid use among older adults in the United States. Arch Intern Med. 2012 Feb 13;172(3):292-3. doi: 10.1001/archinternmed.2011.1408. No abstract available. PMID 22332170
- [Background] Gopinath B, Schneider J, Hartley D, Teber E, McMahon CM, Leeder SR, Mitchell P. Incidence and predictors of hearing aid use and ownership among older adults with hearing loss. Ann Epidemiol. 2011 Jul;21(7):497-506. doi: 10.1016/j.annepidem.2011.03.005. Epub 2011 Apr 21. PMID 21514179
- [Background] Humes LE, Rogers SE, Quigley TM, Main AK, Kinney DL, Herring C. The Effects of Service-Delivery Model and Purchase Price on Hearing-Aid Outcomes in Older Adults: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Am J Audiol. 2017 Mar 1;26(1):53-79. doi: 10.1044/2017_AJA-16-0111. PMID 28252160
- [Background] Lin FR, Niparko JK, Ferrucci L. Hearing loss prevalence in the United States. Arch Intern Med. 2011 Nov 14;171(20):1851-2. doi: 10.1001/archinternmed.2011.506. No abstract available. PMID 22083573
- [Background] Nelson PB, Perry TT, Gregan M, VanTasell D. Self-Adjusted Amplification Parameters Produce Large Between-Subject Variability and Preserve Speech Intelligibility. Trends Hear. 2018 Jan-Dec;22:2331216518798264. doi: 10.1177/2331216518798264. PMID 30191767
- [Background] Urbanski D, Hernandez H, Oleson J, Wu YH. Toward a New Evidence-Based Fitting Paradigm for Over-the-Counter Hearing Aids. Am J Audiol. 2021 Mar 10;30(1):43-66. doi: 10.1044/2020_AJA-20-00085. Epub 2020 Dec 1. PMID 33264578

DOCUMENTS (1):
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT06499805/ICF_000.pdf